CLINICAL TRIAL: NCT03134235
Title: A 4-week Defined, Raw, Plant-based Diet Improves Anthropometric, Hemodynamic, and Other Cardiovascular Risk Factors
Brief Title: Effects of a 4-week Raw, Plant-based Diet on Anthropometric and Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Montgomery Heart & Wellness (Unknown)
Responsible Party: Principal Investigator, Rami Najjar, Student, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19279
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; Elevated Cholesterol; Overweight and Obesity
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Overweight; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Repeated measures, single group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raw, plant-based diet (Experimental): A raw, plant-based diet was prescribed for 4 weeks.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Subjects consumed a raw, vegan diet for 4-weeks with an emphasis on raw fruit and vegetable consumption.

SUMMARY:
This study evaluates the effects of a prescribed 4-week raw, plant-based dietary intervention in the treatment of excess body weight, hypercholesterolemia, and hypertension in the clinical setting.

DETAILED DESCRIPTION:
Plant-based diets have emerged in the literature as effective therapeutic strategies in the reduction of body weight, serum lipids and blood pressure. In addition, raw fruit and vegetable consumption has also been associated with the reduction of these clinical indicators.

Participants were instructed to follow a prescribed, raw, plant-based dietary intervention for four weeks. All animal products, including eggs and dairy, were excluded. Cooked foods, free oils, soda, alcohol and coffee were also to be excluded. All meals and snacks were provided to the participants for the full duration of the intervention. Emphasized were raw fruits and vegetables, while seeds, avocado, raw oats, raw buckwheat, and dehydrated foods were prepared as condiments. Vitamin, herbal, and mineral supplements were to be discontinued unless otherwise clinically indicated. Participants were not advised to alter their exercise habits.

Participants came to a total of 4 follow-up visits. A laboratory panel was obtained at baseline and at 4-weeks. A 24-hour recall was also conducted at baseline and at 4-weeks. Anthropometrics, hemodynamics, and medication needs were assessed on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥25.0 kg/m^2
* Serum low-density lipoprotein cholesterol concentration ≥100
* Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90

Exclusion Criteria:

* Tobacco use
* Drug abuse
* Excessive alcohol consumption (>2 glasses of wine or alcohol equivalent per day for men or >1 glass of wine or alcohol equivalent for woman)
* Current cancer diagnosis
* Estimated glomerular filtration rate <60 mg/dL
* Clinically defined infection
* Mental disability
* Hospitalization <6 months
* Previous exposure to plant-based diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline, follow-up weeks 1-4
  Weight (kg) was documented at baseline and during 4 additional weekly follow-up visits
Change in serum low-density lipoprotein cholesterol (LDL) | Baseline and 4-weeks
  LDL cholesterol (mg/dL) was documented at baseline and after 4-weeks
Change in blood pressure | Baseline, follow-up weeks 1-4
  Systolic and diastolic blood pressure (mmHg) was documented at baseline and during 4 additional weekly follow-up visits

SECONDARY OUTCOMES:
Change in heart rate | Baseline, follow-up weeks 1-4
  Heart rate (beats/min) was documented at baseline and during 4 additional weekly follow-up visits
Change in waist circumference | Baseline, follow-up weeks 1-4
  Waist circumference (cm) was documented at baseline and during 4 additional weekly follow-up visits
Change in serum total cholesterol | Baseline and 4-weeks
  Serum total cholesterol (mg/dL) was documented at baseline and after 4-weeks
Change in serum high-density lipoprotein cholesterol | Baseline and 4-weeks
  Serum HDL (mg/dL) was documented at baseline and after 4-weeks
Change in serum triglycerides | Baseline and 4-weeks
  Triglycerides mg/dL was documented at baseline and after 4-weeks
Change in serum insulin | Baseline and 4-weeks
  Insulin (uU/mL) was documented at baseline and after 4-weeks
Change in serum glucose | Baseline and 4-weeks
  Serum glucose (mg/dL) was documented at baseline and after 4-weeks
Change in serum hemoglobin A1c (HgA1c) | Baseline and 4-weeks
  HgA1c (%) was documented at baseline and after 4-weeks
Change in c-reactive protein (CRP) | Baseline and 4-weeks
  CRP (mg/L) was documented at baseline and after 4-weeks
Change in medication use | Baseline, follow-up weeks 1-4
  Medication needs were assessed weekly

CONTACTS AND LOCATIONS:
Overall Officials: Rami Najjar, Principal Investigator — Texas Woman's University
Locations (1):
- Montgomery Heart & Wellness, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Bazzano LA. Effects of soluble dietary fiber on low-density lipoprotein cholesterol and coronary heart disease risk. Curr Atheroscler Rep. 2008 Dec;10(6):473-7. doi: 10.1007/s11883-008-0074-3. PMID 18937894
- [Background] Bloomer RJ, Kabir MM, Canale RE, Trepanowski JF, Marshall KE, Farney TM, Hammond KG. Effect of a 21 day Daniel Fast on metabolic and cardiovascular disease risk factors in men and women. Lipids Health Dis. 2010 Sep 3;9:94. doi: 10.1186/1476-511X-9-94. PMID 20815907
- [Background] Boeing H, Bechthold A, Bub A, Ellinger S, Haller D, Kroke A, Leschik-Bonnet E, Muller MJ, Oberritter H, Schulze M, Stehle P, Watzl B. Critical review: vegetables and fruit in the prevention of chronic diseases. Eur J Nutr. 2012 Sep;51(6):637-63. doi: 10.1007/s00394-012-0380-y. Epub 2012 Jun 9. PMID 22684631
- [Background] Djousse L, Arnett DK, Coon H, Province MA, Moore LL, Ellison RC. Fruit and vegetable consumption and LDL cholesterol: the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2004 Feb;79(2):213-7. doi: 10.1093/ajcn/79.2.213. PMID 14749225
- [Background] Fraser G, Katuli S, Anousheh R, Knutsen S, Herring P, Fan J. Vegetarian diets and cardiovascular risk factors in black members of the Adventist Health Study-2. Public Health Nutr. 2015 Feb;18(3):537-45. doi: 10.1017/S1368980014000263. Epub 2014 Mar 17. PMID 24636393
- [Background] Jenkins DJ, Kendall CW, Popovich DG, Vidgen E, Mehling CC, Vuksan V, Ransom TP, Rao AV, Rosenberg-Zand R, Tariq N, Corey P, Jones PJ, Raeini M, Story JA, Furumoto EJ, Illingworth DR, Pappu AS, Connelly PW. Effect of a very-high-fiber vegetable, fruit, and nut diet on serum lipids and colonic function. Metabolism. 2001 Apr;50(4):494-503. doi: 10.1053/meta.2001.21037. PMID 11288049
- [Background] Koebnick C, Garcia AL, Dagnelie PC, Strassner C, Lindemans J, Katz N, Leitzmann C, Hoffmann I. Long-term consumption of a raw food diet is associated with favorable serum LDL cholesterol and triglycerides but also with elevated plasma homocysteine and low serum HDL cholesterol in humans. J Nutr. 2005 Oct;135(10):2372-8. doi: 10.1093/jn/135.10.2372. PMID 16177198
- [Background] Le LT, Sabate J. Beyond meatless, the health effects of vegan diets: findings from the Adventist cohorts. Nutrients. 2014 May 27;6(6):2131-47. doi: 10.3390/nu6062131. PMID 24871675
- [Background] Macknin M, Kong T, Weier A, Worley S, Tang AS, Alkhouri N, Golubic M. Plant-based, no-added-fat or American Heart Association diets: impact on cardiovascular risk in obese children with hypercholesterolemia and their parents. J Pediatr. 2015 Apr;166(4):953-9.e1-3. doi: 10.1016/j.jpeds.2014.12.058. Epub 2015 Feb 12. PMID 25684089
- [Background] Mishra S, Xu J, Agarwal U, Gonzales J, Levin S, Barnard ND. A multicenter randomized controlled trial of a plant-based nutrition program to reduce body weight and cardiovascular risk in the corporate setting: the GEICO study. Eur J Clin Nutr. 2013 Jul;67(7):718-24. doi: 10.1038/ejcn.2013.92. Epub 2013 May 22. PMID 23695207
- [Background] Ras RT, Geleijnse JM, Trautwein EA. LDL-cholesterol-lowering effect of plant sterols and stanols across different dose ranges: a meta-analysis of randomised controlled studies. Br J Nutr. 2014 Jul 28;112(2):214-9. doi: 10.1017/S0007114514000750. Epub 2014 Apr 29. PMID 24780090
- [Background] Turner-McGrievy GM, Barnard ND, Scialli AR. A two-year randomized weight loss trial comparing a vegan diet to a more moderate low-fat diet. Obesity (Silver Spring). 2007 Sep;15(9):2276-81. doi: 10.1038/oby.2007.270. PMID 17890496
- [Background] Wu L, Sun D, He Y. Fruit and vegetables consumption and incident hypertension: dose-response meta-analysis of prospective cohort studies. J Hum Hypertens. 2016 Oct;30(10):573-80. doi: 10.1038/jhh.2016.44. Epub 2016 Jun 16. PMID 27306085
- [Background] Yokoyama Y, Nishimura K, Barnard ND, Takegami M, Watanabe M, Sekikawa A, Okamura T, Miyamoto Y. Vegetarian diets and blood pressure: a meta-analysis. JAMA Intern Med. 2014 Apr;174(4):577-87. doi: 10.1001/jamainternmed.2013.14547. PMID 24566947